CLINICAL TRIAL: NCT03919344
Title: Pathophysiological Study of Central Sleep Apnea in Adults With Preserved LVEF
Brief Title: Pathophysiological Study of CSA in Adults With pLVEF
Acronym: PHENOSAX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP 180442
Record Dates: First submitted 2019-03-12; First posted 2019-04-18 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Central Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Central SAS cases (Other): Patients with central apnea
  Interventions: Other: Critical airway closure pressure (Pcrit) measurment; Other: Acoustic pharyngometry; Other: High density surface electroencephalogram neural mapping
- Obstructive SAS controls (Other): Patients with moderate to severe obstructive apnea (apnea-hypopnoea index ≥ 15 / h)
  Interventions: Other: Critical airway closure pressure (Pcrit) measurment; Other: Acoustic pharyngometry
- Snorers controls (Other): Snorers controls : Patients with snoring, with or without mild obstructive apneas (index of apnea-hypopneas <15 / h)
  Interventions: Other: Critical airway closure pressure (Pcrit) measurment; Other: Acoustic pharyngometry

INTERVENTIONS:
Other: Critical airway closure pressure (Pcrit) measurment — Pcrit is measured in awake patient, by applying a gradually decreasing pressure through a nasal NIV mask. Pcrit is defined as the pressure inducing airflow cessation in upper airway
Other: Acoustic pharyngometry — Acoustic pharyngometry will assess the volume of the pharynx and determine if there is an obstacle in the upper airways.
Other: High density surface electroencephalogram neural mapping — Mapping of the respiratory neural network will allow us to study the areas of the brain activated during breathing
  Arms: Central SAS cases

SUMMARY:
Sleep apnea is classically divided into obstructive and central apnea, according to the persistence or otherwise of respiratory movements and the existence or not of pharyngeal collapse during apnea. However, there is evidence to suggest that some mechanisms are common to both types of apnea. Although the pathophysiology of obstructive apnea has been the subject of much work and now seems fairly well known, there is much less data on central apnea. These apneas can occur in different comorbid contexts. They are more frequently present in patients with heart failure, regardless of the etiology, and are associated with an adverse prognosis. The investigators hypothesize that the physiopathology of adult central apnea syndrome involves, in addition to ventilatory control abnormalities, upper airway abnormalities (VAS). The objective is to study the pathophysiology of central SAS, by first comparing the collapse of VAS of central apneic patients to those of patients with simple snoring or obstructive sleep apnea. In a second step, the investigators will analyze the cardiorespiratory coupling and will establish a map of the respiratory neural network in patients with central apnea. The investigators will focus their study on patients with central SAS (with preserved systolic heart function) due to the epidemiology of SAS.

DETAILED DESCRIPTION:
A non-randomized case-control comparative monocentric physiopathology study with 3 parallel groups (one group of cases and two control groups) matched for age and body mass index (individual 1: 1: 1 match), to evaluate changes in the collapse of VAS in central apnea ("central SAS case"), compared to subjects without central apnea ("obstructive SAS" and "single snoring").

Primary objective : Evaluation of changes in upper airway collapse in patients with central sleep apnea syndrome with preserved LVEF heart failure ("central SAS case"), compared with snoring subjects free from sleep apnea syndrome ("Simple snoring witnesses")

Secondary objectives :

* Study the collapsibility of VAS according to the type of apnea ("central SAS case" versus "obstructive SAS case").
* To study the association between the collapsibility of VAS and the global and central apnea-hypopnoea index (IAH).
* Study the association between the type of disorder ("central SAS case" versus "simple snoring controls", "central SAS case" versus "obstructive SAS controls") and cardiorespiratory coupling.
* Study the association between the type of disorder ("central SAS case" versus "simple snoring controls", "central SAS case" versus "obstructive SAS controls") and the CO2 response slope.
* Establish a map of the respiratory neural network in patients with central SAS with preserved ejection fraction.
* Study the association between the volumes in acoustic pharyngometry and the values of the Pcrit

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* Age ≥18 years and ≤85 years
* With preserved LVEF heart failure (defined as LVEF ≥ 45% on ultrasound, MRI or isotopic ventriculography)
* Central SAS Group: Central to severe sleep apnea syndrome, defined by an apnea-hypopnoea index (IAH) greater than 15 per hour, of which at least 30% are central events;
* Obstructive SAS group: Moderate to severe obstructive sleep apnea syndrome, defined by an apnea-hypopnoea index (IAH) greater than 15 per hour, with a central event proportion of less than 30%
* Group "snoring": absence of sleep apnea syndrome or mild sleep apnea syndrome (IAH <15 / h) in polysomnography, and presence of snoring on at least 30% of the night of recording.
* Free, informed and written consent
* Patient affiliated to a social security scheme (beneficiary or beneficiary)

Exclusion Criteria:

* Impossibility of giving the subject informed information
* Participation in a research protocol involving the human person in the previous months if an exclusion directive is given in this protocol
* Use of respiratory or sedative depressant drugs, systemic corticosteroid therapy
* Impaired systolic function (defined by LVEF <45% in ultrasound, MRI or isotopic ventriculography)
* Unstable cardiovascular disease (cardiovascular event of less than one month)
* Recent surgery of the ENT sphere (less than 6 months)
* Central neurological pathology known
* Known, severe respiratory pathology (severity left to the investigator's discretion)
* Renal insufficiency (creatinine clearance <60 mL / min) or severe hepatic impairment
* Primary or secondary hemostasis disorder
* Patient on anticoagulant (antivitamin K, direct oral anticoagulant, heparin and related). Antiplatelet agents are allowed.
* Psychiatric pathology according to DSM-V criteria, unbalanced
* Pulsed saturation with oxyhemoglobin <88% at rest, on awakening
* Allergy to lidocaine
* Patient under tutorship or curatorship
* Failure to perform a prior medical examination
* Tympanic perforation

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Upper airway collapsibility is assessed by Pcrit value in central leep apnea and snoring | 1 day
  Pressure values of VAS (Pcrit) in patients in the "Central SAS" group and in the "Obstructive SAS" group

SECONDARY OUTCOMES:
Upper airway collapsibility is assessed by Pcrit value in central and obstructive sleep apnea | 1 day
  Pcrit value in cm H20 in the obstructive SAS group vs. central SAS group
The association between Pcrit (cm H20) and Apnea-Hypopnoea Index (events/h) | 1 day
  The association between Pcrit (cm H20) and Global and Central Apnea-Hypopnoea Index (events/h)
Chemosensitivity in central sleep apnea is assessed by CO2 response test | 1 day
  CO2 response slope (mL/min/mmHg) in CO2 response test via rebrething method
Cardiorespiratory coupling in central sleep apnea is assessed by RR measurment (mm on EKG) | 1 day
  Parameters of cardiorespiratory coupling to polysomnography
Neural network modifications in sleep apnea are assessed by frequency couplage indice | 1 day
  Respiratory neural network mapping in patients with central SAS with preserved ejection fraction through high density mapping
Volume and collapsibility characteristics in acoustic pharyngometry in the different groups | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pia D'ORTHO, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No